CLINICAL TRIAL: NCT04556331
Title: Brief Online Group Parenting Programme for Anxious Parents of 1-3 Year Olds With the Aim of Reducing Transmission of Anxiety Through Generations: A Feasibility Study
Brief Title: Sowing the Seeds of Confidence: Brief Online Group Parenting Programme for Anxious Parents of 1-3 Year Olds
Acronym: StS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 19/LO/1438 v7 01062020
Record Dates: First submitted 2020-09-07; First posted 2020-09-21 (Actual); Last update posted 2021-02-18 (Actual); Status verified 2020-09

CONDITIONS: Anxiety; Parenting
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Parenting programme (cognitive behavioural) aimed at reducing generational transmission of anxiety — 'Psychoeducation' (psychologically informed information about the topic of transmitting anxiety) and cognitive-behavioural strategies aimed at reducing the transmission of anxiety from parent to young child. These will be shared with a group of maximum 8 remotely delivered, in a didactic format.

SUMMARY:
To pilot a brief group early intervention aimed at reducing or preventing the intergenerational transmission of anxiety, with parents whose child is between 12 and 47 months. To explore feasibility and acceptability of such an intervention with this population.

DETAILED DESCRIPTION:
All participants will attend two group sessions of 'psychoeducation' (psychologically informed information about the topic of transmitting anxiety) and cognitive-behavioural strategies aimed at reducing the transmission of anxiety from parent to young child. The two sessions will be delivered online via Microsoft Teams, last 2 hours each and will run one week apart. Outcome and acceptability measures will be collected before, immediately after, and 6 weeks after the intervention. Feasibility data (e.g. drop-out rate) will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* current or recent (within 2 years) primary diagnosis of anxiety disorder or self-report of clinically impairing anxiety problem within last 2 years,
* parent of child aged 12-47 months at time of intervention,
* access to an internet connection and smart phone/computer will be required to take part,
* male or female,
* resident in England,
* and over the age of 18

Exclusion Criteria:

* current severe co-morbid diagnoses, e.g. psychosis or acute suicidal risk (as the nature of the intervention is brief and in a group, the level of support needed to keep those with severe mental health disorders safe will not be available),
* current alcohol or drugs misuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-09-25 (Actual); Primary Completion 2021-01-20 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Number of participants who consented to take part as percentage of those who expressed initial interest. | Total across recruitment period (up to 11 weeks, October 2020 to mid December 2020)
  Percentage of count (people consent to take part / people expressing interest in response to advertising). To indicate feasibility of larger trial.
Actual attendance at each session as percentage of expected attendance | Total across intervention period (up to 9 weeks, mid October 2020 to mid December 2020)
  Percentage of count (people scheduled to attend each session / people who actually attended). To indicate feasibility of larger trial.
Number of participants who provided completed questionnaire measures | Total across intervention and 6 week follow-up period (up to 15 weeks, mid October 2020 to January 2021)
  Percentage of recruited participants who completed questionnaire measures at each of the three collection timepoints.
Acceptability of Intervention Measure (AIM) and Intervention Appropriateness Measure (IAM) (Weiner, Lewis et al. 2017) | Collected twice: immediately after intervention attendance (same day) and after 6 weeks.
  Validated measure of acceptability of an intervention - Acceptability of Intervention Measure (AIM) and Intervention Appropriateness Measure (IAM) (Weiner, Lewis et al. 2017)
Open text questions about participants' views on the acceptability | Collected twice: immediately after intervention attendance (same day) and after 6 weeks.
  Open text questions to gather qualitative information about participants' perspectives on usefulness, accessibility and unintended negative consequences

SECONDARY OUTCOMES:
Change in score on Brief Infant Toddler Social and Emotional Assessment (Briggs-Gowan, Carter et al. 2002) | Collected three times to access change: Before intervention, immediately after end of intervention (same day) and 6 weeks after.
  Parent report measure of child social, emotional and behavioural difficulties. This is a 42-item parent-report screening tool validated with parents of children aged 12 to 47 months. Maximum score is 84 and minimum score is 0. The higher the score the worse the outcome.
Change in score on Depression Anxiety Stress Scale (Henry and Crawford 2005) | Collected three times to access change: Before intervention, immediately after end of intervention (same day) and 6 weeks after.
  Parent report questionnaire measure of stress, anxiety and depression in parents. This is a 21-item scale. The minimum score is 0 and the maximum score is 63, higher score is a worse outcome.
Bespoke questionnaire about self-reported use and confidence in behaviours specifically targeted in intervention. | Collected three times to access change: Before intervention, immediately after end of intervention (same day) and 6 weeks after.
  Bespoke questionnaire about 8 specific parenting behaviours targeted in the intervention, each rated on a 5-point Likert scale (4 are reverse scored). Minimum score is 0 and maximum score is 40. The higher the score the 'worse' the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Fiona Challacombe, PhD DClinPsy, Principal Investigator — King's College London
Locations (1):
- South London and Maudsley NHS Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Palmer E, Woolgar M, Carter B, Cartwright-Hatton S, Challacombe FL. Preventing anxiety in the children of anxious parents - feasibility of a brief, online, group intervention for parents of one- to three-year-olds. Child Adolesc Ment Health. 2023 Feb;28(1):33-41. doi: 10.1111/camh.12596. Epub 2022 Aug 18. PMID 35983606